CLINICAL TRIAL: NCT00243360
Title: Optimizing Antibiotic Use in Long Term Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: U18HS011113-01 (AHRQ)
Record Dates: First submitted 2005-10-21; First posted 2005-10-24 (Estimated); Last update posted 2005-10-24 (Estimated); Status verified 2005-10

CONDITIONS: Urinary Tract Infection, Antibiotic Use
Keywords: Urinary tract infections,; antibiotic use,; long term care facilities
MeSH Terms: conditions — Urinary Tract Infections

INTERVENTIONS:
Behavioral: diagnostic and treatment clinical algorithms

SUMMARY:
The purpose of this study was to determine if a multi-faceted intervention to implement diagnostic and therapeutic algorithms for management of suspected urinary infection in nursing home residents could reduce antibiotic prescribing for urinary indications in this population.

DETAILED DESCRIPTION:
Antibiotic use is intense in nursing homes and frequently inappropriate when prescribed for urinary indications. Evidence from randomized controlled trials suggests that treatment of asymptomatic bacteriuria, the presence of bacteria in the urine in the absence of urinary symptoms, is not beneficial. Despite this, one in three prescriptions for urinary indications are for asymptomatic bacteriuria. To improve antibiotic prescribing in this setting we conducted a cluster randomized trial of a strategy to implement diagnostic and treatment algorithms for urinary infection. 24 nursing homes were randomized to either the intervention (implemented at the nursing home level using a multi-faceted approach: small group interactive sessions for nurses, one-on-one interviews for physicians, videotapes, written material, and outreach visits) or to usual care.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals- all residents eligible
2. Nursing homes

   * Free standing long term care facilities with >100 beds
   * No stated policy for diagnosis or treatment of urinary tract infections
   * The facility agrees to refrain from introducing new strategies for antibiotic utilization or clinical pathways during study

Exclusion Criteria:

-

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-01; Study Completion 2003-07

PRIMARY OUTCOMES:
Antimicrobial prescriptions

SECONDARY OUTCOMES:
Urinary cultures,
hospitalizations, deaths

CONTACTS AND LOCATIONS:
Overall Officials: Mark B Loeb, MD MSc FRCPC, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada